CLINICAL TRIAL: NCT06510764
Title: A Randomized Controlled Trial of Ziyin-Xiehuo Chinese Medicine Herbs Combined With Intradermal Acupuncture for the Treatment of Girl's Idiopathic Precocious Puberty With Yin Deficiency and Fire Hyperactivity
Brief Title: A Trial of Chinese Traditional Medicine Combining With Intradermal Acupuncture for Treating Precocious Puberty
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23Y11921100
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Precocious Puberty; Treatment; Alternative Medicine; Acupuncture
MeSH Terms: conditions — Puberty, Precocious | interventions — Medicine, Chinese Traditional

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Chinese Medicine+acupuncture (Experimental): Subjects in this group will be treated with traditional Chinese medicine and intradermal acupuncture point stimulation for 6 months.
  Interventions: Other: intradermal needles; Drug: Ziyinxiehuo Granules of traditional Chinese Medicine
- Traditional Chinese Medicine (Active Comparator): Subjects in this group will be treated withTraditional Chinese Medicine for 6 months.
  Interventions: Drug: Ziyinxiehuo Granules of traditional Chinese Medicine

INTERVENTIONS:
Other: intradermal needles — Disposable intradermal needles will be used for acupoint stimulation and Tai Chong, Taixi, Sanyinjiao, Hegu as well as Yanglingquan are chosen for acupuncture point. Acupuncture point pressure will last for 10 minutes each time, three times per day, and the intradermal needles will be changed every 2 days.
  Arms: Traditional Chinese Medicine+acupuncture
Drug: Ziyinxiehuo Granules of traditional Chinese Medicine — Ziyinxiehuo Granules of traditional Chinese Medicine which includes shengdi 15g, xuanshen 9g, zexie 9g, zhimu9g, huangbai 9g, zhiguiban 9g, maiya 15g, tiandong 9g, zhigancao 9g,and will be administered after dissolved, 1package every time, 2 times per day after a meal.
  Other Names: traditional Chinese Medicine for nourishing Yin and purging fire

SUMMARY:
A randomized controlled study will be conducted to evaluate the therapeutic effect of traditional Chinese medicine and acupoints stimulation on children with idiopathic precocious puberty.

DETAILED DESCRIPTION:
Traditional Chinese medicine is effective for precocious puberty which is mild or moderate, but not effective for the one that is severe and rapidly progressing. Acupuncture can effectively regulate sex hormone levels and ovarian function, promote ovulation, and have therapeutic effect for polycystic ovary syndrome and irregular menstruation. Studies have shown that acupuncture and auricular point compression stimulation is effective for premature thelarche, yet there are few studies on idiopathic precocious puberty. Clinical evidence is still needed to support whether acupuncture point stimulation combined with traditional Chinese Medicine herbs can enhance the effect and prevent the progression into severe or rapidly progressing precocious puberty, hence the study is to be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Girls are diagnosed as Idiopathic precocious puberty, and their age of onset ≤7.5years;
* Tanner stages of breast in female patients ≤ Tanner III stage, diameters of mammillary nucleus ≤ 3cm; •B-type ultrasonography: the volume of uterus≥ 3ml, the volume of ovary≥1.5ml, the diameter of follicle≥4mm;
* Bone age: compared the chronological age, the bone age is less than 1 year and the bone age <10 years old;
* No GnRH analogs or Sex hormones were administrated in the past; and All above are needed at the same time.

Exclusion Criteria:

* Precocity caused by the central nervous system organic diseases;
* Precocious precocity caused by congenital hypothyroidism, congenital adrenal hyperplasia, adrenal tumor and ovarian or testicular neoplasms as well as McCune-Albright syndrome, etc;
* Precocious precocity with a family history of diseases such as tumor, leukemia, diabetes, systemic lupus erythematous;
* Pseudo sexual precocity and partial precocious puberty.

Ages: 4 Years to 9 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 170 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
The percentage of subjects' mammary nucleus minification or disappearance at the third month. | from baseline to the third month.
  The diameters of mammary nucleus will be measured with rulers along the median line of the breast at baseline,the third month and the sixth month. The subject numbers of mammary nucleus minification or disappearance at third month will be recorded. The percentage=the subject numbers of mammary nucleus minification or disappearance /total subject numbers in this group ×100%.

SECONDARY OUTCOMES:
the change in bone age／the change in chronological age after six months | from baseline to the sixth month
  The bone age will be measured with X-ray and evaluated with G-P Atlas method at baseline and the sixth month. the change in bone age= bone age after six months-bone age at baseline, the change in chronological age is six months.

CONTACTS AND LOCATIONS:
Overall Officials: Sun Yanyan, Master, Principal Investigator — Children's Hospital of Fudan University
Locations (2):
- China (2):
  - Children's Hospital of Fudan university, Shanghai, Shanghai Municipality
  - Children's Hospital of Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No